CLINICAL TRIAL: NCT07262879
Title: Effect of Nurse-Led Intradialytic Stretching Exercises on Muscle Cramp Burden Among Patients Undergoing Maintenance Hemodialysis: A Randomized Controlled Trial
Brief Title: Stretching Exercises for Dialysis Patients to Reduce Muscle Cramps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ahmed Mostafa Shehata, Lecturer of Medical Surgical Nursing, faculty of Nursing, Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC/01092024/Ali
Record Dates: First submitted 2025-11-20; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Muscle Cramp; Renal Dialysis; Exercise Therapy; Nursing Care
Keywords: Nurse-led intervention; Intradialytic stretching; Hemodialysis symptoms; Muscle cramps; Exercise therapy; Non-pharmacological intervention; Symptom management; Proactive nursing care
MeSH Terms: conditions — Muscle Cramp

STUDY DESIGN:
Intervention Model Description: The study describes a "parallel-group randomized controlled trial" where participants were randomized into one of two distinct groups that received different interventions concurrently (study group vs. control group) for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (nurse-led intradialytic stretching exercises) (Experimental): This arm received a structured, nurse-led lower-limb stretching program in addition to their usual hemodialysis (HD) care. The intervention was designed to be a proactive, non-pharmacological strategy to prevent intradialytic muscle cramps.
  Interventions: Other: Nurse-Led Intradialytic Stretching Exercises
- The control group (usual care) (No Intervention): This control arm received routine hemodialysis care without any structured exercise program.

INTERVENTIONS:
Other: Nurse-Led Intradialytic Stretching Exercises — Participants in the intervention group received a nurse-led, supervised intradialytic lower-limb stretching program. The standardized protocol was administered during the first 1-2 hours of hemodialysis sessions, twice a week, for a total of 15 sessions over approximately 8 weeks. The protocol consisted of four stretches targeting major lower-limb muscle groups: ankle dorsiflexion, gastrocnemius stretch, soleus stretch, and hamstring stretch. Each stretch was held for 20-30 seconds and repeated three times per limb. HD nurses, trained in the protocol and vascular access safety, delivered the intervention. Adherence and correct technique were monitored and documented for each session using a structured fidelity checklist.
  Arms: The intervention group (nurse-led intradialytic stretching exercises)

SUMMARY:
This single-center, parallel-group randomized controlled trial aims to evaluate the effect of a nurse-led intradialytic stretching program on the burden of muscle cramps in patients receiving maintenance hemodialysis (HD). Sixty adult patients on thrice-weekly HD with a history of lower-limb cramps will be randomized 1:1 to either an intervention group or a usual care control group.

The intervention consists of a standardized protocol of supervised lower-limb stretches (ankle dorsiflexion, gastrocnemius, soleus, and hamstring stretches). Each stretch will be held for 20-30 seconds and repeated three times per limb. The protocol will be delivered by HD nurses during dialysis sessions, twice a week for a total of 15 sessions over approximately eight weeks. Fidelity will be monitored using a structured checklist. The control group will receive routine care without structured exercises.

The primary outcome is the post-intervention cramp intensity category, measured using the Arabic Muscle Cramp Severity and Characteristics Questionnaire (MC-SCQ). Secondary outcomes include cramp frequency, duration, pain intensity, leg temperature perception, and discomfort/functional interference.

DETAILED DESCRIPTION:
1. The Problem: The Burden of Intradialytic Muscle Cramps For patients undergoing maintenance hemodialysis (HD), the treatment is a life-sustaining necessity that comes with a significant symptom burden. Among the most common and disruptive of these symptoms are intradialytic muscle cramps-sudden, involuntary, and painful muscle contractions, primarily in the lower limbs. These episodes are not merely a minor inconvenience; they represent a serious clinical challenge. Cramps can be severe enough to forcibly halt a dialysis session, trigger distress calls to nurses, and necessitate urgent interventions such as sterile saline boluses or adjustments to the ultrafiltration rate. These reactive measures disrupt the dialysis process, can lead to hemodynamic instability, and increase nursing workload. For the patient, the experience is one of pain, anxiety, and a diminished quality of life. Estimates suggest these cramps affect a wide proportion, between 20% to 85%, of the chronic HD population.
2. The Proposed Solution: A Proactive, Nurse-Led Intervention Traditional management of these cramps has largely been reactionary. This study proposes to test a paradigm shift: moving from reactive treatment to proactive, nurse-led prevention. The intervention under investigation is a standardized protocol of lower-limb stretching exercises, administered during the dialysis session (intradialytically). The rationale is grounded in exercise physiology: sustained stretching is believed to improve muscle flexibility, enhance local circulation, and modulate neuromuscular excitability, potentially raising the threshold at which a cramp is triggered. By leveraging the time patients are already connected to the dialysis machine and the constant presence of a nurse, this strategy offers a low-cost, non-pharmacological, and patient-centric approach that aligns with nursing values of health promotion and continuity of care.
3. Study Design and Rigor

   To generate high-quality evidence, this study employs a single-center, parallel-group, randomized controlled trial (RCT) design. In this design, 60 eligible adult patients from the Beni-Suef University Hospital HD unit will be randomly assigned to one of two groups:

   The Intervention Group: Will receive the nurse-led intradialytic stretching program in addition to usual care.

   The Control Group: Will continue to receive usual care without any structured exercise program.

   This randomization process is intended to ensure that the groups are similar in all key aspects at the beginning of the study. To safeguard the integrity of the intervention, the research team will use a fidelity checklist to ensure every stretching session is delivered consistently and correctly.
4. The Intervention in Detail The stretching protocol is designed to be both effective and feasible within a busy dialysis unit. It targets the primary muscle groups involved in cramps: the ankle dorsiflexors, gastrocnemius, soleus, and hamstrings.

   Execution: During the first 1-2 hours of their dialysis session, patients in the intervention group will perform a series of supervised stretches. Each stretch will be held for 20-30 seconds and repeated three times for each limb.

   Safety: A paramount concern is patient safety, particularly regarding the vascular access site. Nurses will be trained to ensure all stretches are performed away from the access arm, with no compromise to needle security or tubing.

   Dosage: The program will be administered twice a week for approximately eight weeks, totaling 15 supervised sessions.
5. Measuring the Impact

The effect of the stretching program will be measured using the Arabic Muscle Cramp Severity and Characteristics Questionnaire (MC-SCQ). This tool is designed to capture the multi-dimensional burden of cramps by assessing:

Frequency of episodes Duration of cramps Pain Intensity Functional Interference and discomfort Leg Temperature Perception

Assessments will be conducted at baseline and at the end of the 8-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 21 years or older.
* Undergoing maintenance hemodialysis on a thrice-weekly schedule.
* Have been on hemodialysis for at least 3 months.
* Clinically stable.
* Have a history of intradialytic lower-limb muscle cramps in the preceding month.
* Able to provide informed consent.

Exclusion Criteria:

* Musculoskeletal or neurological disorders that limit safe lower-limb stretching.
* Femoral vascular access or recent lower-limb vascular procedures.
* Undergoing their first or an emergency hemodialysis session.
* Inability to provide informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Post-intervention muscle cramp intensity category | 8 weeks
  Post-intervention muscle cramp intensity category, as measured by the Arabic Muscle Cramp Severity and Characteristics Questionnaire (MC-SCQ). The total MC-SCQ score (range 0-13) was mapped into a four-level ordinal categorical variable: None (0), Mild (1-4), Moderate (5-8), or Severe (9-13). The distribution of participants across these categories was compared between the study and control groups at the end of the 8-week intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Baseline Characteristics: Age, sex, comorbidities, hemodialysis vintage, and baseline physiological parameters (e.g., blood pressure, calcium levels).
  Primary Outcome Data: Individual post-intervention cramp intensity category scores (None, Mild, Moderate, Severe) from the Arabic MC-SCQ questionnaire.
  Secondary Outcome Data: De-identified scores for all MC-SCQ sub-domains, including:
  Cramp frequency
  Cramp duration
  Pain intensity
  Discomfort/functional interference
  Leg temperature perception
  Intervention Data: Session-level adherence and fidelity checklist scores for participants in the intervention arm.
  This data will be stripped of all direct identifiers (e.g., name, medical record number) to protect participant confidentiality.
Supporting Information: Study Protocol, SAP
Time Frame: Start Date: The IPD and supporting information will become available 3 months after the main results of the clinical trial are accepted for publication.
  End Date: The data will be made available for a period of 5 years from the start date.
Access Criteria: Who can access:
  Researchers, including graduate students and investigators from academic institutions, healthcare organizations, and non-profit entities.
  Access will be granted to those with a methodologically sound proposal for use in achieving the goals outlined in their approved proposal.
  What they can access:
  Individual Participant Data (IPD): De-identified dataset including baseline characteristics, primary outcome (cramp intensity category), and all secondary outcomes (frequency, duration, pain, etc.).
  Supporting Information: The full Study Protocol and Statistical Analysis Plan (SAP).
  How they can access it:
  Mechanism: Data and documents will be shared via a secure file transfer service or a trusted data repository link upon approved request.
  Process: Interested parties must submit a formal request via email to the corresponding author (Ahmed Mostafa).
  Oversight: Requests will be reviewed by the study's principal investigators to ensure scientific validity & ethical approval.

REFERENCES:
- [Background] Takahashi A. The pathophysiology of leg cramping during dialysis and the use of carnitine in its treatment. Physiol Rep. 2021 Nov;9(21):e15114. doi: 10.14814/phy2.15114. PMID 34762357
- [Background] Soliman AR, Soliman KM, Abdelaziz TS, Ahmed RM, Abdellatif DA, Darwish RA, Abosaif N, Maamoun H, Hammad H, Zayed B, Fayed A, Abdelhamid YM, El-Khashab SO, Elkhatib M. The evolution of nephrology practice in Egypt: legacy, current challenges, and future directions-a narrative review. Ren Fail. 2025 Dec;47(1):2509784. doi: 10.1080/0886022X.2025.2509784. Epub 2025 May 29. PMID 40438027
- [Background] Sasirekha, C. (2017). Effectiveness of Intradialytic Stretching Exercise on Muscle Cramps among Patients Undergoing Haemodialysis at Selected Hospitals, Salem (Doctoral dissertation, Sri Gokulam College of Nursing, Salem).
- [Background] Romeu-Perales M, Segura-Orti E, Cana-Poyatos A, Toquero-Correa M, Benavent-Caballer V, Pans-Alcaina D, Garcia-Maset R, Garcia-Testal A. The Effect of Intradialytic Exercise Using Virtual Reality on the Body Composition of Patients with Chronic Kidney Disease. Nutrients. 2024 Jun 20;16(12):1968. doi: 10.3390/nu16121968. PMID 38931320
- [Background] Miller KC, McDermott BP, Yeargin SW, Fiol A, Schwellnus MP. An Evidence-Based Review of the Pathophysiology, Treatment, and Prevention of Exercise-Associated Muscle Cramps. J Athl Train. 2022 Jan 1;57(1):5-15. doi: 10.4085/1062-6050-0696.20. PMID 34185846
- [Background] Miller KC, Burne JA. Golgi tendon organ reflex inhibition following manually applied acute static stretching. J Sports Sci. 2014;32(15):1491-7. doi: 10.1080/02640414.2014.899708. Epub 2014 Apr 9. PMID 24716521
- [Background] Kot G, Wrobel A, Kuna K, Makowka A, Nowicki M. The Effect of Muscle Cramps During Hemodialysis on Quality of Life and Habitual Physical Activity. Medicina (Kaunas). 2024 Dec 18;60(12):2075. doi: 10.3390/medicina60122075. PMID 39768954
- [Background] Kimmel PL, Varela MP, Peterson RA, Weihs KL, Simmens SJ, Alleyne S, Amarashinge A, Mishkin GJ, Cruz I, Veis JH. Interdialytic weight gain and survival in hemodialysis patients: effects of duration of ESRD and diabetes mellitus. Kidney Int. 2000 Mar;57(3):1141-51. doi: 10.1046/j.1523-1755.2000.00941.x. PMID 10720966
- [Background] Hargrove N, El Tobgy N, Zhou O, Pinder M, Plant B, Askin N, Bieber L, Collister D, Whitlock R, Tangri N, Bohm C. Effect of Aerobic Exercise on Dialysis-Related Symptoms in Individuals Undergoing Maintenance Hemodialysis: A Systematic Review and Meta-Analysis of Clinical Trials. Clin J Am Soc Nephrol. 2021 Apr 7;16(4):560-574. doi: 10.2215/CJN.15080920. Epub 2021 Mar 25. PMID 33766925
- [Background] Gelfman R, Ingraham BS, Sandhu GS, Lerman A, Lewis B, Gulati R, Pellikka PA, Higgins SD, Singh M. Stretching to Reduce Pain-Related Disability Among Echocardiographic and Interventional Laboratory Employees-A Pilot Study. J Soc Cardiovasc Angiogr Interv. 2024 May 2;3(5):101353. doi: 10.1016/j.jscai.2024.101353. eCollection 2024 May. PMID 39132460
- [Background] Alvarez L, Brown D, Hu D, Chertow GM, Vassalotti JA, Prichard S. Intradialytic Symptoms and Recovery Time in Patients on Thrice-Weekly In-Center Hemodialysis: A Cross-sectional Online Survey. Kidney Med. 2019 Dec 20;2(2):125-130. doi: 10.1016/j.xkme.2019.10.010. eCollection 2020 Mar-Apr. PMID 32734233
- [Background] Alshammari B, Edison JS, Alkubati SA, Alrasheeday AM, Albagawi B, Alharbi LL, Motakef HI, Alshammari L, Siam BGAE, Alharbi NA, Assiri W, Almoqad AA, Aldibas AI, Alshammari F. Effectiveness of exercise in reducing symptom burden among hemodialysis patients: a non-pharmacological intervention approach. Front Public Health. 2025 Jul 9;13:1580689. doi: 10.3389/fpubh.2025.1580689. eCollection 2025. PMID 40703153